CLINICAL TRIAL: NCT05180370
Title: Questionnaire-based Multicenter Prospective Observational Study Evaluating Patient Perception, Compliance and Adaptation in the Management of Heart Failure - ADAPTATION HF
Brief Title: Multicenter Prospective Observational Study Evaluating the Management of Heart Failure
Acronym: ADAPTATION-HF
Status: Completed | Type: Observational
Sponsor: AstraZeneca Turkey (Industry)
Collaborators: Klinar CRO (Other)
Responsible Party: Sponsor
Other Study IDs: K-J019
Record Dates: First submitted 2021-09-03; First posted 2022-01-06 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Questionnaire; ECHO; Prospective; Cross-Sectional
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatient or inpatient diagnosed with Heart Failure at least 6 months ago: ADAPTATION HF is a prospective, observational, cross-sectional, multicenter, survey-based study. Patients who applied to the cardiology outpatient clinic with a preliminary diagnosis of HF or were hospitalized for HF and had a diagnosis of HF for at least 6 months will be included in the study.
  Interventions: Other: Questionnaies

INTERVENTIONS:
Other: Questionnaies — Data entry staff who will be assigned to the centers for 2 weeks will apply a questionnaire consisting of different questions to the patients referred to them by clinicians with the diagnosis of HF (presented in the appendix to this protocol). In addition, Pittsburg Sleep Quality Index will be applied to all cases.

SUMMARY:
ADAPTATION HF is a prospective, observational, cross-sectional, multicenter, survey-based study. Patients who applied to the cardiology outpatient clinic with a preliminary diagnosis of HF or were hospitalized for HF and had a diagnosis of HF for at least 6 months will be included in the study.

DETAILED DESCRIPTION:
ADAPTATION HF is a prospective, observational, cross-sectional, multicenter, survey-based study. Patients who applied to the cardiology outpatient clinic with a preliminary diagnosis of HF or were hospitalized for HF and had a diagnosis of HF for at least 6 months will be included in the study. Data entry staff who will be assigned to the centers for 2 weeks will apply a questionnaire consisting of different questions to the patients referred to them by clinicians with the diagnosis of HF. In addition, Pittsburg Sleep Quality Index will be applied to all cases. In addition, clinical features of HF from the current file of the cases (NYHA, comorbid conditions, comorbid diseases, blood pressure, heart rate, last drugs used, latest biochemistry (BNP/NTproBNP if available), hematology test results, most recent ECG , most recent echocardiography, coronary angiography report, if available) will be recorded. No additional examination/procedure will be performed for the study, only the data of the examinations requested by the clinician in routine clinical practice will be entered. A total of 500 patients from 10 centers will be included in this study over a six-month period.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient or inpatient diagnosed with Heart Failure at least 6 months ago
* Male or female patient aged 18 and over
* Signed written informed consent form

Exclusion Criteria:

* newly diagnosed heart failure
* CRY requiring dialysis
* Serious liver and lung disease
* LVAD/heart transplantation
* HF due to possible temporary cause (myocarditis, peripartum CMP in the first 6 months, takotsubo etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases admitted to the cardiology outpatient clinic or hospitalized for Heart Failure and diagnosed with HF for at least 6 months will be included in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
General Status of the patients | 6 months
  At the end of the six-month recruitment period, demographic, symptoms, clinical follow-up status, disease information, treatment compliance, and awareness assessment will be performed on all included patients.

SECONDARY OUTCOMES:
HF Risk Factors | 6 Months
HF Percutaneous Intervention History & Operation History | 6 Months
Medications Used for HF | 6 Months
HF Comorbidities | 6 Months
HF ECHO Results | 6 Months
HF Laboratory Results | 6 Months

CONTACTS AND LOCATIONS:
Locations (10):
- Turkey (Türkiye) (10):
  - Ankara City Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Eskişehir Osmangazi University Medical Faculty, Eskişehir
  - Başkent University Istanbul Health Practice and Research Center Hospital, Istanbul
  - Dr. Siyami Ersek Chest Cardiac and Vascular Surgery T&R Hospital, Istanbul
  - Istanbul University - Cerrahpaşa, Cardiology Institute, Istanbul
  - Dokuz Eylül University Medical Faculty, Izmir
  - Ege University Medical Faculty, Izmir
  - Tepecik Training and Research Hospital, Izmir
  - Mersin University Medical Faculty, Mersin

IPD SHARING:
Plan to Share IPD: No